CLINICAL TRIAL: NCT07183358
Title: Effect of Family-Supervised Multimodal Prehabilitation Throughout Preoperative Neoadjuvant Chemotherapy on Clinical Outcomes in Gastric Cancer Patients: A Single-Center Randomized Controlled Trial
Brief Title: Family-Supervised Prehabilitation to Reduce Postoperative Complications After Neoadjuvant Chemotherapy in Gastric Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Zhou Yanbing, Chief Physician, Affiliated Hospital of Qingdao University, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QYFYEC2025-156
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Stomach Neoplasms; Neoadjuvant Therapy
Keywords: prehabilitation; postoperative complications; multimodal; family-supervised; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms; Postoperative Complications | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Standard Care Only) (Active Comparator): Participants in this arm will receive standard neoadjuvant chemotherapy followed by radical gastrectomy, along with standard ERAS (Enhanced Recovery After Surgery) perioperative management. No prehabilitation intervention will be provided.
  Interventions: Other: Standard Care
- Prehabilitation + Standard Care (Experimental): Participants will receive a family-supervised multimodal prehabilitation program throughout the neoadjuvant chemotherapy period until the day before surgery. The intervention includes personalized nutritional support, home-based exercise training, and psychological counseling, in addition to standard neoadjuvant chemotherapy, surgery, and ERAS management.
  Interventions: Behavioral: Family-supervised Multimodal Prehabilitation

INTERVENTIONS:
Behavioral: Family-supervised Multimodal Prehabilitation — A comprehensive prehabilitation program initiated at the start of neoadjuvant chemotherapy and continued until the day before surgery. The intervention includes:
  1. Nutritional support: individualized dietary counseling and supplementation plans supervised by clinical nutritionists;
  2. Exercise training: home-based aerobic and resistance exercises monitored via wearable devices and weekly video/phone follow-ups;
  3. Psychological support: structured counseling sessions to reduce anxiety, improve treatment adherence, and enhance quality of life.
  Family members are trained to assist with supervision and compliance. The total duration is approximately 10-16 weeks, depending on the chemotherapy schedule.
  Arms: Prehabilitation + Standard Care
Other: Standard Care — Standard neoadjuvant chemotherapy followed by radical gastrectomy with standard ERAS-based perioperative management, without any additional prehabilitation intervention. Participants receive routine nutritional, nursing and medical care according to hospital guidelines. The aim is to maintain current clinical practice as the control condition for comparison with the experimental prehabilitation program.
  Arms: Control Group (Standard Care Only)

SUMMARY:
This study evaluates whether a family-supervised exercise-nutrition-psychology program can reduce complications after stomach-cancer surgery. Eligible patients are adults who will receive chemotherapy before surgery. Participants are randomly assigned to either the multimodal prehabilitation program plus usual care or usual care alone. The main outcome is the rate of serious complications within 30 days after surgery. Potential benefits include fewer complications and faster recovery; risks are minimal and mainly related to mild exercise fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Histologically proven gastric adenocarcinoma by gastroscopy
* Clinical stage T2-4a, N any, M0 planned for neoadjuvant chemotherapy plus radical gastrectomy
* ECOG performance status 0-1; ASA class I-III
* Able to understand the study and provide signed informed consent

Exclusion Criteria:

* Previous or concurrent malignancies
* Emergent conditions (bleeding, perforation, obstruction) requiring immediate surgery
* Pregnant or lactating women
* Severe psychiatric disorders
* Prior major abdominal surgery (except laparoscopic cholecystectomy)
* Unstable angina, myocardial infarction, or cerebrovascular event within 6 months
* Continuous use of NSAIDs, corticosteroids, or probiotics within 1 month
* Simultaneous surgery for other diseases
* FEV1 < 50 % predicted
* Any condition that, in the investigator's opinion, contraindicates participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative complications within 30 days after surgery | Within 30 days after surgery
  Postoperative complications include surgical site infection, anastomotic leakage, bleeding, pneumonia, urinary tract infection, and other surgery-related adverse events occurring within 30 days after radical gastrectomy.

SECONDARY OUTCOMES:
Intestinal barrier function indicators (Claudin-1, Occludin, ZO-1 expression) | Baseline, before surgery, and postoperative day 7
  Expression levels of tight junction proteins in intestinal mucosa, measured by immunohistochemistry or Western blot.
Nutritional status (serum albumin, prealbumin, transferrin, hemoglobin, body weight) | Baseline, before surgery, and postoperative day 7
  Assessment of nutritional markers and body weight changes during treatment.
Karnofsky Performance Status (KPS) score | Baseline, before surgery, and postoperative day 7
  A standardized measure of functional ability and general health status.
Intraoperative blood loss and operative time | Day of surgery
  Total intraoperative blood loss (mL) and duration of surgery (minutes).
Length of postoperative hospital stay | Up to 30 days after surgery
  Number of days from surgery to hospital discharge.
Disease-free survival (DFS) at 6 months and 1 year | 6 months and 1 year after surgery
  Time from surgery to recurrence or death from any cause.
Biological barrier: gut microbiota composition and diversity | Baseline, before surgery, and postoperative day 7
  Fecal samples will be analyzed using 16S rRNA gene sequencing to evaluate microbial diversity and composition as indicators of the biological barrier.
Chemical barrier: fecal MUC2 protein level and goblet cell density | Baseline, before surgery, and postoperative day 7
  Fecal MUC2 concentration measured by ELISA and goblet cell density in small intestinal mucosa assessed by histopathological staining.
Immune barrier: fecal sIgA level and mucosal T-cell counts (CD3⁺, CD4⁺, CD8⁺) | Baseline, before surgery, and postoperative day 7
  Fecal secretory IgA (sIgA) measured by ELISA; mucosal CD3⁺, CD4⁺, and CD8⁺ T-cell densities evaluated by immunohistochemistry.

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao University Affiliated Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Golder HJ, Papalois V. Enhanced Recovery after Surgery: History, Key Advancements and Developments in Transplant Surgery. J Clin Med. 2021 Apr 12;10(8):1634. doi: 10.3390/jcm10081634. PMID 33921433
- [Background] Fleurent-Gregoire C, Burgess N, McIsaac DI, Chevalier S, Fiore JF Jr, Carli F, Levett D, Moore J, Grocott MP, Copeland R, Edbrooke L, Engel D, Testa GD, Denehy L, Gillis C. Towards a common definition of surgical prehabilitation: a scoping review of randomised trials. Br J Anaesth. 2024 Aug;133(2):305-315. doi: 10.1016/j.bja.2024.02.035. Epub 2024 Apr 26. PMID 38677949
- [Background] Biondi A, Lirosi MC, D'Ugo D, Fico V, Ricci R, Santullo F, Rizzuto A, Cananzi FC, Persiani R. Neo-adjuvant chemo(radio)therapy in gastric cancer: Current status and future perspectives. World J Gastrointest Oncol. 2015 Dec 15;7(12):389-400. doi: 10.4251/wjgo.v7.i12.389. PMID 26690252
- [Background] Kang, Y.-K., Yook, J. H., Park, Y.-K., et al. (2019). Phase III randomized study of neoadjuvant chemotherapy (CT) with docetaxel (D), oxaliplatin (O) and S-1 (S) (DOS) followed by surgery and adjuvant S-1, vs surgery and adjuvant S-1, for resectable advanced gastric cancer (GC) (PRODIGY). Annals of Oncology, 30(10), 1637-1645.
- [Background] Newton AD, Datta J, Loaiza-Bonilla A, Karakousis GC, Roses RE. Neoadjuvant therapy for gastric cancer: current evidence and future directions. J Gastrointest Oncol. 2015 Oct;6(5):534-43. doi: 10.3978/j.issn.2078-6891.2015.047. PMID 26487948
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593